CLINICAL TRIAL: NCT05231317
Title: Effect of the Sustainable Diet on Gut Microbiota and the Metabolome: a Randomised Crossover Study
Acronym: SUSUGUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Fondazione Edmund Mach (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: REC/20/0008
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Microbiota; Nutrition, Healthy
Keywords: Plant-based diet; Western diet; Gut microbiota,; Trimethylamine N-oxide; Human intervention study.
MeSH Terms: interventions — Diet, Plant-Based; Diet, Western

STUDY DESIGN:
Intervention Model Description: Cross-over single-blinded
Who Masked: Participant
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Plant-based diet (Experimental): Diet rich in fruit and vegetables (42% carbohydrates, 17.2% fibres; 15% proteins and 43% fats).
  Interventions: Other: Plant-based diet
- Active Comparator: Western diet (Active Comparator): Diet Rich in Processed Foods (48% carbohydrates, 10.4% fibres; 14% proteins and 39% fats).
  Interventions: Other: Western diet

INTERVENTIONS:
Other: Plant-based diet — 16 days with all foods provided
  Arms: Experimental: Plant-based diet
Other: Western diet — 16 days with all foods provided
  Arms: Active Comparator: Western diet

SUMMARY:
Unhealthy diets are closely linked to non-communicable diseases and constitute higher risk of morbidity and mortality than unsafe sex, alcohol, tobacco and drugs use combined. According to the World Health Organization (WHO), a healthy diet follows a plant-based pattern with low quantities of red meat and a low simple sugar intake. It would also reduce anthropological ecologic impact. We hypothesize that a plant-based diet will beneficially modify the gut microbiota and metabolome, influencing also Trimethylamine N-oxide (TMAO), a metabolite associated to CVD.

This study has a randomized single blind crossover design that compares a plant-based diet towards a control western diet. It is applied to volunteers aged 18-70 years, N=20. Each dietary intervention (plant-based and western) would last for 16 consecutive days separated by a minimum of 7 weeks washout period (intervention 1-washout-intervention 2). Samples of blood urine and faeces will be collected at day 1 and 14 of each intervention. On day 14 will be performed L-carnitine challenge with 1200mg of L-carnitine to test the levels of TMAO), in for the next 2 consecutive days (24h and 48h post treatment).

ELIGIBILITY:
Inclusion Criteria:

* Free-living, apparently healthy adults
* Bmi>18
* Aged 18-70 years at recruitment
* Non-smokers

Exclusion criteria:

* Non-free-living adults
* Adults <18 or >70 years at recruitment
* BMI<18
* Current smokers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Gut microbiota changes | Change over 14 days
  Significant changes in the number of bifidobacteria
Quantification of Trimethylamine N-oxide | Day 16
  Changes in response to L-Carnitine challenge

SECONDARY OUTCOMES:
Bioactivity of faecal water | Change over 14 days
  Measured by using faecal water as basis for growth media (ex vivo measure)
Effects on inflammatory markers of both diets | Change over 14 days
  Cytokine analysis via ELISA test (MagPix)
Ex vivo effects of faecal water on gut pathobionts | Day 14
  Co-culturing the aqueous phase of faeces with C. difficile to assess changes in its biology
Quantification of phytochemicals | Change over 14 days
  Measured by LC-MS
Quantification of Short Chain Fatty Acids (SCFA) | Change over 14 days
  Measured by nuclear magnetic resonance (NMR)

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, Londonderry, United Kingdom